CLINICAL TRIAL: NCT07118189
Title: Laying the Foundation for Building a Resilient KPNC Community in the Face of Worsening Air Quality Due to Wildfire Smoke
Acronym: DS-F
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Laura Myers, Principal Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2293325
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Exacerbation of COPD; Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease (COPD); air pollution; wildfire smoke
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N95 Respirators

STUDY DESIGN:
Intervention Model Description: randomized in-home intervention pilot trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: data analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who are randomized into the intervention will receive N95 masks to be worn outdoors and an indoor air cleaner in the room that the participant spends the most time in their home. Both intervention and control arms will receive education.
  Interventions: Device: N95 masks and indoor air cleaner
- Control (No Intervention): Both intervention and control arms will receive education.

INTERVENTIONS:
Device: N95 masks and indoor air cleaner — Participants who are randomized into the intervention will receive N95 masks to be worn outdoors and an indoor air cleaner in the room that the participant spends the most time in their home. Both intervention and control arms will receive education.
  Arms: Intervention

SUMMARY:
The overarching goal of this project is to conduct a pilot intervention in high-risk Kaiser Permanente Northern California patients with chronic obstructive pulmonary disease to mitigate their exposure to poor air quality and decrease exacerbations of lung disease.

DETAILED DESCRIPTION:
Over the past decade, the frequency and impact of wildfires has steadily worsened across California, a trend that is expected to continue as climate change becomes an urgent, everyday reality. This means that the number of Kaiser Permanente Northern California (KPNC) members exposed to unhealthy air quality due to wildfire smoke will increase dramatically. Unsurprisingly, vulnerable patients are disproportionately impacted, such as those with chronic obstructive pulmonary disease (COPD). In this rigorous pilot, we will deploy a pilot in-home intervention to non-smoking, oxygen-dependent patients who have frequent exacerbations of COPD to mitigate their exposure to poor air quality and reduce exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* KPNC patients
* enrolled in Care Plus
* non-smoking
* oxygen-dependent
* adults aged ≥65 years old
* have had membership for at least 1 year prior to data extraction not counting </=3mo gaps)
* have known COPD (at least 2 encounters with COPD ICD codes over a 3 year period in the 10 years prior to data extraction using the following ICD codes: ICD-9 491.21, 491.22, 491.8, 491.9, 492.8, 493.2, 493.21, 493.22, 496 and ICD-10 J44.1, J44.0, J41.8, J44.9, J42)15
* have picked up at least 1 controller inhaler at the pharmacy within 1 year prior to data extraction
* at least 2 exacerbations of COPD treated in any setting (outpatient or acute care) within 1 year before to data extraction.

Exclusion Criteria:

* with <1 year of continuous membership prior to the date they entered the cohort, allowing for 3-month, non-contiguous gaps
* any diagnosis with any of the past or present problems: blindness, dementia, deaf or hearing impaired, hospice admission, "tracheostomy" procedure code or problems and/or attached to a ventilator
* hearing, visually, physically, memory, and/or speech impaired
* those on the "Do Not Call" list
* non-English speakers.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
feasibility (by percent of enrolled patients who complete all follow-up assessments) | 30 days
  % of enrolled patients who complete all follow-up assessments
fidelity | 30 days
  electrical sensors on the air cleaners showing the device was on for >80% of follow-up time

SECONDARY OUTCOMES:
average screen-to-enrollment ratio | Through study completion, an average of 18 months
  how many patients were contacted to enroll 1 patient
indoor and outdoor PM2.5 concentrations | 30 days
  air quality monitoring devices inside and outside the home, which record data internally when not connected to the internet
respiratory quality of life | 30 days
  via St George's respiratory questionnaire for COPD - Part 1 : Symptoms component (frequency & severity) with a 1-month recall; Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall (dichotomous (true/false) except last question (4-point Likert scale)); Scores range from 0 to 100, with higher scores indicating more limitations
effectiveness | 30 days
  FEV1 improvement by portable spirometry
acceptability | 30 days
  >90% reporting satisfied/very satisfied on 5-point Likert scale as well as in qualitative interviews for feedback about the intervention, specifically which aspect of the intervention was most/least helpful and most/least burdensome, including aspects that should be changed to increase participation in future trials
Urine oxidative stress | 30 days
  analysis of urinary F2-isoprostanes and Specific Gravity (SG)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northern California Division of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No
organizational guidance